CLINICAL TRIAL: NCT00445354
Title: A Randomized Controlled Clinical Trial Comparing the Effect of 1g of Daily Cinnamon Plus Usual Care to Usual Cre on the Hemoglobin A1c of Uncontrolled Type 2 Diabetics
Brief Title: Randomized Controlled Clinical Trial of Cinnamon to Lower Hemoglobin A1c
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eglin AFB Regional Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20060194H
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Diabetes
Keywords: cinnamon; diabetes; hemoglobin a1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cinnamon

SUMMARY:
This study will randomize diabetics with hemoglobin A1c greater than 7.0 to receive either cinnamon plus usual care or usual care alone. Hemoglobin A1c will be measured at intake and after 90 days.

DETAILED DESCRIPTION:
As the worldwide incidence of diabetes increases, the search for dietary adjuncts to treat this life-altering disease becomes far ranging. Cinnamon is purported to be a natural insulin sensitizer without any known adverse events. Both in vitro and in vivo animal studies have shown that cinnamon is an insulin sensitizer1. Several compounds within cinnamon have been identified as possible sources of this sensitization process.

To-date, three small randomized trials studying cinnamon in human diabetics have been published. Khan et al. reported that fasting serum glucose could be reduced by 18-29% after 40 days of supplementation with 1, 3, or 6 g of cinnamon (Cinnamomum cassia) in type 2 diabetics. 2 This study had several limitations that included failure to measure hemoglobin A1C, all patients were Pakistani, and no power analysis was documented. Vanschoonbeek, et al.3 report a small RCT of postmenopausal women with well-controlled type 2 diabetes which showed no change in HbA1C or fasting glucose. Once again no power analysis is reported. Mang et al. 4 conducted a RCT of type 2 diabetics treated with aqueous extract of cinnamon for 4 months. They report a 15% decrease in fasting glucose and no change in HbA1C over the duration of this trial. Subjects had HbA1C less than 7% and again no power analysis was included in this study.

This study will address whether cinnamon at the dose of 1g daily in addition to usual care lowers hemoglobin A1c compared to usual care. Power analysis indicates that 63 per group are needed and we will recruit 70 patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics greater tahn 18 years of age

Exclusion Criteria:

* allergy to cinnamon pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c

SECONDARY OUTCOMES:
diabetes medications

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Principal Investigator — Eglin AFB Hospital
Locations (1):
- Eglin AFB Regional Hospital, Eglin Air Force Base, Florida, United States

REFERENCES:
- [Background] Talpur N, Echard B, Ingram C, Bagchi D, Preuss H. Effects of a novel formulation of essential oils on glucose-insulin metabolism in diabetic and hypertensive rats: a pilot study. Diabetes Obes Metab. 2005 Mar;7(2):193-9. doi: 10.1111/j.1463-1326.2004.00386.x. PMID 15715893
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804
- [Background] Vanschoonbeek K, Thomassen BJ, Senden JM, Wodzig WK, van Loon LJ. Cinnamon supplementation does not improve glycemic control in postmenopausal type 2 diabetes patients. J Nutr. 2006 Apr;136(4):977-80. doi: 10.1093/jn/136.4.977. PMID 16549460
- [Background] Mang B, Wolters M, Schmitt B, Kelb K, Lichtinghagen R, Stichtenoth DO, Hahn A. Effects of a cinnamon extract on plasma glucose, HbA, and serum lipids in diabetes mellitus type 2. Eur J Clin Invest. 2006 May;36(5):340-4. doi: 10.1111/j.1365-2362.2006.01629.x. PMID 16634838
- [Derived] Crawford P. Effectiveness of cinnamon for lowering hemoglobin A1C in patients with type 2 diabetes: a randomized, controlled trial. J Am Board Fam Med. 2009 Sep-Oct;22(5):507-12. doi: 10.3122/jabfm.2009.05.080093. PMID 19734396